CLINICAL TRIAL: NCT03211429
Title: Randomized Clinical Trial Evaluating the Effectiveness of Three Interventions Programs to Improve Functionality and Decrease Fear of Falling in the Elderly
Brief Title: Effectiveness of Three Interventions to Reduce Fear of Falling and Improve Functionality in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Caldas (Other)
Collaborators: Universidad de Manizales (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1386316
Record Dates: First submitted 2017-01-16; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Fear of Falling
MeSH Terms: interventions — Cognitive Behavioral Therapy; Tai Ji

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive behavioural therapy (Active Comparator): The program aims to teach participants how to deal with their concerns about falls and related avoidance of activity, in order to increase their physical, social and functional activities. The cognitive behavioural intervention program, provides by psychologists, consists of eight group sessions, 60 minutes each. During each session a main theme is addressed. The themes of the program are: concerns about falls; thoughts about falling; physical exercise; asserting oneself; overcoming personal barriers; safe behaviour; and managing concerns about falls.
  Interventions: Behavioral: Cognitive behavioural therapy
- Tai chi (Active Comparator): Subjects in the Tai Chi group undertook supervised Tai Chi training in the Yang style of 24 movements, for one hour, once a week for 8 weeks. The first 5 min was allocated for warm-up, with the rest of the time for Tai Chi practice.
  Interventions: Other: Tai chi
- Postural control exercise (Active Comparator): Individually adjusted progressive and specific postural control training, provided by physiotherapists for one hour, one time per week for 8 weeks. The exercise is progressive and specific to functional postural control tasks. It comprises elements that represent activities included in, and required for, independent daily living, such as maintaining balance when sitting, standing and walking; and also reacting to loss of balance.
  Interventions: Other: Postural control exercise

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — The program aims to teach participants how to deal with their concerns about falls and related avoidance of activity
  Arms: Cognitive behavioural therapy
Other: Tai chi — Tai Chi training in the Yang style of 24 movement
  Arms: Tai chi
Other: Postural control exercise — Individually adjusted progressive and specific postural control training,
  Arms: Postural control exercise

SUMMARY:
Fear of falling is a major health problem among community-dwelling older adults that may contribute to avoidance of activities that they are capable of performing. Studies show that the fear of falling may lead to a continual, complex decline in older adults that includes a loss of auto efficacy, restriction of physical activities and social participation, physical frailty, falls and disability. Apart from these effects, the fear of falling may also have financial implications for health care systems and the general public. Several interventions have been shown to reduce fear of falling with multifactorial interventions, including physical and behavioral components, being most successful. Behavioral components usually comprise strategies to reduce catastrophic thinking and fear-related avoidance behaviors while physical components usually comprise falls prevention exercise programs. However, multifactorial programs are not always feasible or preferred by older people. In this framework, the objective of this works is to assess the effects (benefits and effectiveness) of three interventions programs (Tai Chi, postural control exercises and behavioral therapy intervention) to improve functionality and decrease fear of falling in older people living in the community.

DETAILED DESCRIPTION:
Fear of falling is common among elderly people. Fear of falling can be associated with reductions in physical and social activities and negative impacts on quality of life. Several interventions have been shown to reduce the fear of falling, but their effectiveness has not been compared. The objective of this study is to evaluate the effectiveness of three interventions programs to improve functionality and decrease fear of falling in the Elderly. Effective interventions to lessen fear of falling could therefore have significant consequences for individuals, their families and healthcare delivery systems.

Methods/Design: This is a controlled, randomized clinical trial of individual assignment, carried out on community living elderly, from Manizales (Colombia) who reporting fear of falling with restriction of activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older people
* People who reported fear of falling
* "Leganés Cognitive Test" ≥23
* SPPB ≤ 9

Exclusion Criteria:

* Some cognitive affection and/or medical condition that may affect the intervention
* Permanent use of wheelchair
* People who have received prior protocolized management for fear of falling

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Fear of falling | Prospective change from baseline to end of intervention (8 weeks)
  Fear of falling is evaluated using Falls Efficacy Scale International questionnaire
Functional mobility | Prospective change from baseline to end of intervention (8 weeks)
  Functional mobility is evaluated using gait speed and Short Physical performance Battery (SPPB).

SECONDARY OUTCOMES:
Falls | Prospective change from baseline to end of intervention (8 weeks)
  Number of falls in the last year evaluated by open question to the participant
Depression | Prospective change from baseline to end of intervention (8 weeks)
  Prospective change from baseline to end of intervention (8 weeks) as measured by the scale of Yesavage
Handgrip | Prospective change from baseline to end of intervention (8 weeks)
  Prospective change from baseline to end of intervention (8 weeks) Measured through the dynamometer
Daily life activities | Prospective change from baseline to end of intervention (8 weeks)
  Daily life activities at the instrumental level measured through the Lawton and Brody scale
Self-Rated Health | Prospective change from baseline to end of intervention (8 weeks)
  Subjective assessment of health status by simple dichotomous scale and ordinal scale (Likert scale) with 5 options
Postural control | Prospective change from baseline to end of intervention (8 weeks)
  under reduced or conflicting sensory conditions and fall risk were investigated, using the Biodex Balance System

CONTACTS AND LOCATIONS:
Overall Officials: Carmen L Curcio, Principal Investigator — Universidad de Caldas
Locations (1):
- Universidad de caldas, Manizales, Caldas Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available after publication of results. Data will be shared to interested researchers who are planning to perform a meta-analysis. They should write an email to the main contact explaining what type of analysis they will perform and what data they require from the study. Only those data that are considered relevant for the analysis will be shared. Researchers who receive the data should be committed to safeguarding them and complying with and protecting copyright

REFERENCES:
- [Derived] Duenas EP, Ramirez LP, Ponce E, Curcio CL. [Effect on fear of falling and functionality of three intervention programs. A randomised clinical trial]. Rev Esp Geriatr Gerontol. 2019 Mar-Apr;54(2):68-74. doi: 10.1016/j.regg.2018.09.013. Epub 2018 Nov 24. Spanish. PMID 30482460